CLINICAL TRIAL: NCT02726113
Title: Vitamin D and Prostate Cancer: A Randomized Clinical Study
Brief Title: Vitamin D and Prostate Cancer: A Clinical Study Enrolling Subjects Undergoing Prostatectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: MUSC Pro# 12772
Record Dates: First submitted 2011-12-06; First posted 2016-04-01 (Estimated); Results first posted 2019-12-03 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-12

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; vitamin D
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention: Cholecalciferol (Active Comparator): vitamin D3 (cholecalciferol) supplementation at 4000 IU daily for approximately two months prior to surgery (prostatectomy).
  Interventions: Drug: cholecalciferol
- Placebo (Placebo Comparator): softgel (containing no active ingredient) daily for approximately two months prior to surgery (prostatectomy).
  Interventions: Other: placebo

INTERVENTIONS:
Drug: cholecalciferol — softgels 4000 IU daily for approximately two months prior to surgery (prostatectomy).
  Other Names: vitamin D3
  Arms: Intervention: Cholecalciferol
Other: placebo — softgel containing no active ingredient daily for approximately two months prior to surgery (prostatectomy).
  Arms: Placebo

SUMMARY:
The study population will be 80 adult men who have been diagnosed with prostate cancer who are scheduled to have their prostate surgically removed at either the Medical University of South Carolina (MUSC) or the Ralph H. Johnson VAMC, both located in Charleston, SC. The men will be randomized into two groups: one group will take vitamin D3 supplementation and the other will take a placebo. Blood levels of vitamin D3 will be obtained at the beginning of the study and again after two months, just prior to the surgical procedure (prostatectomy). Prostate tissue will be obtained from the surgical procedure and studied for the effect of vitamin D on the prostate cancer cells.

DETAILED DESCRIPTION:
This study will enroll 80 (40 per study arm) subjects (>18 years of age), recently diagnosed with prostate cancer (histologically documented adenocarcinoma of the prostate), who are scheduled to undergo prostatectomy.

Eligible subjects will be recruited in the Urology Clinic at MUSC or Ralph H. Johnson VAMC. All subjects will be refered to the study by their Urologist. At the baseline visit, consent will be obtained before any study procedures are initiated. A blood sample will be obtained for 25(OH)D3 analysis. Subjects will be randomized to either the intervention group (vitamin D3 4000 IU daily) or the placebo group and take the study medication for approximately two months before their scheduled prostatectomy. The final study visit is the day of surgery. A blood sample for 25(OH)D3 analysis will be obtained. Prostate tissue will be collected from the Pathologist for (a) genomics (RNA sequencing) analysis; (b) proteomics (proteins, glycons and lipids) analysis and (c) Vitamin D Receptor (VDR) by immunohistochemistry.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of prostate cancer (by prostate biopsy)
* Scheduled to undergo a prostatectomy
* Ability to give his own consent to participate in the study

Exclusion Criteria:

* Serum 25(OH)D level less than 8ng/ml or greater than 50 ng/ml
* Vitamin D3 supplementation greater than or equal to 1000 IU daily

Ages: 19 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-10; Primary Completion 2015-03 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sebastiano Gattoni-Celli, MD, Principal Investigator — MUSC Department of Radiation Oncology
Locations (2):
- United States (2):
  - Ralph H. Johnson VA Medical Center, Charleston, South Carolina
  - MUSC (Medical University of South Carolina), Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects with diagnosed prostate cancer, who were scheduled for prostatectomy, were randomized into D3 supplementation vs Placebo groups prior to surgey
Pre-assignment Details: Overall Study
Groups:
- Intervention: vitamin D3 (cholecalciferol) supplementation at 4000 IU daily for approximately two months prior to surgery (prostatectomy).
Period: Total Enrollment
Arm/Group | Intervention | Placebo
Started | 28 | 22
Completed | 24 | 19
Not Completed | 4 | 3
Not completed — Physician Decision | 0 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Insurance non-coverage for surgery | 1 | 1
Period: Genomic Analysis
Arm/Group | Intervention | Placebo
Started | 19 | 14
Completed | 15 | 12
Not Completed | 4 | 2
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Insurance non-coverage for surgery | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Placebo | Total
Number analyzed (Participants) | 28 | 22 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 17 | 34
  >=65 years | 11 | 5 | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 28 | 22 | 50
Race/Ethnicity, Customized [Number; unit: participants]
  African American | 10 | 10 | 20
  Caucasian/Non-Hispanic | 18 | 12 | 30
Region of Enrollment [Number; unit: participants]
  United States | 28 | 22 | 50

OUTCOME MEASURES:

1. Primary Outcome: Changes in Serum Levels of Vitamin D [25(OH)D3] in Subjects in the Supplementation Group and Those in the Control Group (Placebo).
Description: Baseline vitamin D3 levels will be obtained at enrollment and approximately two months later during the surgical procedure (prostatectomy). These D3 levels will be evaluated for the 27 participants who had genomic analysis and compared by race (Caucasian and AA).
Time Frame: approximately two months from baseline to date of prostatectomy (exit)
Population: 27 participants, who had genomic analysis (RNA sequencing), were evlauated for their serum level of D3 at baseline and exit. Intervention: 9 Caucasian/5 AA and Control: 8 Caucasian/5 AA
Measure: Mean (Full Range); unit: ng/ml
Groups:
- Control: Placebo softgel (containing no active ingredient) daily for approximately two months prior to surgery (prostatectomy).
Arm/Group | Intervention | Control
Number analyzed (Participants) | 14 | 13
ng/ml
  Baseline Caucasian: number analyzed (Participants) | 9 | 8
  Baseline Caucasian | 29.8 [11.7 to 46.9] | 34.8 [21.3 to 56.9]
  Exit Caucasian: number analyzed (Participants) | 9 | 8
  Exit Caucasian | 46.94 [35.0 to 70.8] | 29.6 [19.3 to 41.8]
  Baseline AA: number analyzed (Participants) | 5 | 5
  Baseline AA | 21.66 [14.1 to 30.3] | 26.06 [15.6 to 33.7]
  Exit AA: number analyzed (Participants) | 5 | 5
  Exit AA | 48.84 [32.8 to 69.7] | 24.88 [18.4 to 34.1]

2. Secondary Outcome: Number of Gene Transcripts Identified Regulated by Vitamin D Supplementation in Both AA and European American Participants
Description: The intent of this outcome measure was to identify the number of gene transcripts found to be differentially expressed (where a difference or change has occurred) in both AA and EA subjects upon vitamin D supplementation. The transcripts differentially expressed were compared to the transcripts in the "Placebo" Arm/Group.
Time Frame: up to 8 months post prostatectomy
Population: All study participants completed genomic analysis
Measure: Number; unit: differentially expressed transcripts
Units Other Than Participants: Total transcripts
Groups:
- All Study Participants: All study participants undergoing genomic analysis of prostrate tissue
Arm/Group | All Study Participants
Number analyzed (Participants) | 27
Number analyzed (Total transcripts) | 8237
differentially expressed transcripts | 346

ADVERSE EVENTS:
Time Frame: two months, or the period of each subject's participation
Description: Each participant was questionned by a study team member whether he had experienced any adverse or unanticipated events from time of enrollment to just prior to his prostatectomy. Each participant's health record was reviewed from date of enrollment to date of prostatectomy (exit).
Arm/Group | Intervention | Placebo
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/22
Other Adverse Events (participants affected / at risk) | 0/28 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No